CLINICAL TRIAL: NCT02950571
Title: A Randomized Controlled Trial Examining the Effectiveness of Digital Picture Frame Use on the Long Term Inpatient Experience
Brief Title: RCT Examining the Effectiveness of Digital Picture Frame Use in Inpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Sean Kidd, Independent Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 074/2016
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia; Psychosis; Psychosis NOS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Routine care is comprised of a high level of support from an interdisciplinary team with access to unit-specific and centralized programming
  Interventions: Behavioral: Standard Care
- Digital Picture Frames (Experimental): Setup: Over 1-2, approximately 30 minute meetings pictures will be uploaded onto the device from picture files provided by the participant and/or their family or an open online source (e.g., Google Images) that are relevant and of interest to the participant.
  Installation: The picture frames are secured to a surface in the participant's room (most typically a table) by facilities staff. Participants are instructed in its use.
  Check in: At midpoint (2 weeks) an RA will check in with the participant to informally discuss whether or not it continues to work, is being used, and if they want more pictures uploaded. If the latter is requested step 1 will be repeated.
  Interventions: Behavioral: Digital Picture Frame

INTERVENTIONS:
Behavioral: Digital Picture Frame — The intervention is the provision of digital picture frames in long stay inpatient rooms in a ward at CAMH.
  Arms: Digital Picture Frames
Behavioral: Standard Care — High level of support from an interdisciplinary team.
  Arms: Standard Care

SUMMARY:
This study will be a randomized controlled trial that investigates the effectiveness of digital picture frames (DPF) installed in inpatient rooms on long stay inpatient wards servicing schizophrenia clients at CAMH. The effects on client experience will consider the domains of self-concept, interactions with healthcare staff, perception of space, and implications for the recovery process. The comparison of inpatient client experience with DPFs versus a control group (Treatment as Usual - TAU), offers the opportunity to examine the effectiveness of this type of environmental adaptation. This trial builds upon earlier work that demonstrated the feasibility of DPFs in this context.

DETAILED DESCRIPTION:
Long term stays in mental health facilities have been shown to have unique challenges and implications. To a considerable extent these challenges grow out of the stigmatized nature of severe mental illnesses (SMI) such as schizophrenia. The social and self-stigma surrounding SMI can have major effects on those affected including decreased self-esteem, self-deprecation, and the development of a self-concept defined by the illness. When stigmatized interpretations of mental illness are internalized, those affected can find it very challenging to sustain non-illness identities and can ultimately result in the loss of non-illness related aspects of self-concept. Inpatient contexts are particularly challenging in this regard, with non-illness oriented identities very difficult to sustain given considerations of power differentials with providers, the reduction of autonomy and choice, and the removal of the individual from environments that are demonstrative of non-illness aspects of self.

Accordingly, a randomized controlled trial design will be used to consider the question: Does having a DPF in psychiatric inpatient unit rooms lead to improvements in interactions with the clinical team, perceptions of enhanced quality of physical space, and an improvement in the sustaining of non-illness aspects of self-concept? While the promising feasibility study findings might suggest hypotheses of improvement in these domains, we will consider this study exploratory given the complex environments inpatient units represent in the study of care quality and outcomes and the modest scope of this intervention. Finally, we will continue to collect feasibility data qualitatively, to inform further refinement of metrics and otherwise consider enhancements in intervention and research design.

ELIGIBILITY:
Inclusion Criteria:

* All participants will have severe mental illness (SMI) defined as diagnosis with a major mental illness (in practice, will be primarily schizophrenia spectrum) and inherent to hospital admission will be substantive contact with services and disability affecting day-to-day functioning (Ruggeri, Leese, Thornicroft, Bisoffi, & Michelle, 2000).
* Admitted to a CAMH inpatient unit, specifically units 2-2 and 2-3, with an anticipated length of stay of 4 weeks or more, as determined by the clinical team
* Chart diagnosis of a major mental illness
* Determined appropriate for study by staff psychiatrist and clinical team (capacity to consent confirmed, no precautions against having the device in the participant's room indicated)
* 18 years of age or older
* Proficiency in English

Exclusion Criteria:

* Do not meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Recovery Self Assessment (RSA; O'Connell et al., 2005) | Baseline and after 4 weeks (post intervention)
  To examine the degree to which inpatient staff are perceived as recognizing the individuality of the individual and engage in a hopeful and holistic manner. 4 items from the patient version will be used (1-5 point Likert scale).
Client Satisfaction Questionnaire-8 (CSQ-8; Attkisson et al., 1995) | After 4 weeks (post intervention)
  Investigators will only use the general satisfaction question from this measure (1-5 point Likert scale). Only participants in the intervention arm will complete this question.
Change in Empowerment Scale (Rogers et al., 1997) | Baseline and after 4 weeks (post intervention)
  Measures dimensions of self efficacy, self stigma and self concept (1-9 point Likert scale).
Change in Modified Engulfment Scale (McCay & Seeman, 1998) | Baseline and after 4 weeks (post intervention)
  Only two items from this measure focussing specifically on self-concept will be used (1-5 point Likert scale).
Change in Rosenberg Self-Esteem Scale (Rosenberg, 1965) | Baseline and after 4 weeks (post intervention)
  The broadest reaching and high factor loading item, 'On the whole I am satisfied with myself' will be used (1-4 point Likert scale).
Change in Scale to Assess Therapeutic Relationship (STAR; Mcguire-Snieckus et al., 2007) | Baseline and after 4 weeks (post intervention)
  Three items assessing common factors in the therapeutic relationship with the clinical team are from the scale will be used (1-5 point Likert scale).
Change in Satisfaction with the physical environment of the inpatient unit | Baseline and after 4 weeks (post intervention)
  One question developed my investigators due to lack of standardized measures to specifically measure participant satisfaction with the physical environment of the inpatient unit (1-5 point Likert scale)
Change in Satisfaction with the rooms on the inpatient unit | Baseline and after 4 weeks (post intervention)
  One question developed by investigators due to lack of standardized measures to specifically measure participant satisfaction with their room on the inpatient unit (1-5 point Likert scale)
Semi structured interviews | After 4 weeks (post intervention)
  SC participants will be asked broad questions about how satisfied they were with the inpatient unit space and what might be improved. These same questions will be asked of DPF participants, but will be followed by questions specific to the DPF support.

CONTACTS AND LOCATIONS:
Overall Officials: Sean A Kidd, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Connell M, Tondora J, Croog G, Evans A, Davidson L. From rhetoric to routine: assessing perceptions of recovery-oriented practices in a state mental health and addiction system. Psychiatr Rehabil J. 2005 Spring;28(4):378-86. doi: 10.2975/28.2005.378.386. PMID 15895922
- [Background] Attkisson, C. C., & Greenfield, T. K. (1995). The Client Satisfaction Questionnaire (CSQ) scales. Outcome assessment in clinical practice. Baltimore, MD: Williams & Wilkins, 2-10.
- [Background] Rogers ES, Chamberlin J, Ellison ML, Crean T. A consumer-constructed scale to measure empowerment among users of mental health services. Psychiatr Serv. 1997 Aug;48(8):1042-7. doi: 10.1176/ps.48.8.1042. PMID 9255837
- [Background] McCay EA, Seeman MV. A scale to measure the impact of a schizophrenic illness on an individual's self-concept. Arch Psychiatr Nurs. 1998 Feb;12(1):41-9. doi: 10.1016/s0883-9417(98)80007-1. PMID 9489173
- [Background] Rosenberg, M. (1965). Rosenberg self-esteem scale (RSE). Acceptance and commitment therapy. Measures package, 61.
- [Background] McGuire-Snieckus R, McCabe R, Catty J, Hansson L, Priebe S. A new scale to assess the therapeutic relationship in community mental health care: STAR. Psychol Med. 2007 Jan;37(1):85-95. doi: 10.1017/S0033291706009299. Epub 2006 Nov 9. PMID 17094819
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addictions teachings hospital. — http://www.camh.ca/en/research/Pages/research.aspx